CLINICAL TRIAL: NCT06178419
Title: Safety and Efficacy of Remote Ischemic Conditioning for Cerebral Ischemia in Patients With Takayasu Arteritis: a Prospective Cohort Study
Brief Title: Remote Ischemic Conditioning for Cerebral Ischemia in Patients With Takayasu Arteritis (TARIC-1)
Acronym: TARIC-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, ZHAO YI, MD, Professor, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TARIC-1
Record Dates: First submitted 2023-11-21; First posted 2023-12-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cerebral Ischemia; Takayasu Arteritis
Keywords: Cerebral Ischemia; Takayasu Arteritis; remote ischemic conditioning
MeSH Terms: conditions — Brain Ischemia; Takayasu Arteritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): The RIC protocol includes five cycles of 5-min inflation to 200mmHg and 5-min deflation.
  Interventions: Device: RIC
- sham RIC group (Sham Comparator): The sham RIC protocol includes five cycles of 5-min inflation to 60mmHg and 5-min deflation.
  Interventions: Device: sham-RIC

INTERVENTIONS:
Device: RIC — RIC is a non-invasive therapy that is performed by automated pneumatic cuffs placed on unilateral arms. The RIC protocol includes five cycles of 5-min inflation to 200mmHg and 5-min deflation.
  Arms: RIC group
Device: sham-RIC — Sham-RIC is a non-invasive therapy that is performed by automated pneumatic cuffs placed on unilateral arms. The sham RIC protocol includes five cycles of 5-min inflation to 60mmHg and 5-min deflation.
  Arms: sham RIC group

SUMMARY:
The aim of this study is to evaluate the safety and efficacy of remote ischemic conditioning ( RIC ) in the protection of cerebral ischemia in patients with Takayasu arteritis ( TAK ). The study was designed as a prospective, double-blind, exploratory randomized controlled study. The entire study included a screening period and a treatment observation period ( a total of 24 weeks ). All patients with cerebral ischemia of TAK will be randomly divided into RIC group and sham RIC group at 1:1 ratio. On the basis of receiving the conventional drug therapy, the patients will be treated with RIC or sham RIC treatment twice daily for six month. The clinical data of patients at baseline and each follow-up will be collected, including basic information, disease activity assessment, laboratory indicators, imaging indicators, treatment data, adverse events, etc.The Primary outcome is the mean cerebral blood flow improvement rate ( mCBF-IR ) of TAK patients after 24 weeks-treatment. Secondary endpoints include the incidence of major adverse cerebrovascular events ( MACE ) , the change value of arterial transit time ( ATT ) in pCASL hypoperfusion area compared with baseline, occurrence of RIC-related adverse reactions, the changes of hematological indexes and disease activity score, etc. This study will provide insights into the preliminary proof of principle, safety, and efficacy of RIC in cerebral ischemia in patients with Takayasu arteritis ( TAK ), and this data will provide parameters for future larger scale clinical trials if efficacious.

DETAILED DESCRIPTION:
Clinical symptoms, routine follow-up laboratory tests, other serological indicators (VEGF, NGF, ET-1, ACE), PAF, PDGF, etc.), vascular involvement, cranial MRI, vascular injury score, disease activity and treatment will be collected at baseline. After RIC or sham RIC intervention, clinical symptoms, laboratory tests, disease activity, treatment and RIC-related adverse reactions will be collected at 1m, 2m,3m and 6m. the data of vascular involvement, cranial MRI, vascular injury score and disease activity will also be collected at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled the 1990 American College of Rheumatology Classification Criteria for TAK
* Inactive state
* Male and female, aged 18-65 years old
* The presence of supra-aortic vascular involvement ( including but not limited to the left and right sides of the common carotid artery, subclavian artery, vertebral artery involvement )
* Decreased cerebral blood perfusion in the whole brain ( compared with healthy people ) or local ( left and right brain contrast ) suggested by pseudo-Continuous arterial spin labeling ( pCASL ) -MRI
* Voluntary participation in this study, signed informed consent

Exclusion Criteria:

* Complications that endanger the function of important organs, such as uncontrollable heart failure, severe heart valve disease, severe hypertension, severe myocardial ischemia, pulmonary hypertension, acute cerebral infarction, arterial dissection or aneurysm rupture, etc
* There are serious complications, such as poorly controlled diabetes, renal insufficiency, cardiopulmonary insufficiency, mental illness or malignant tumor
* There were moderate to severe stenosis of brachial artery in both upper limbs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Mean cerebral blood flow improvement rate | during baseline to 6 months after therapy
  Mean cerebral blood flow improvement rate ( mCBF-IR ) of TAK patients will be obtained by pseudo-continuous arterial spin labeling ( pCASL ) -MRI.

SECONDARY OUTCOMES:
Incidence of major adverse cerebrovascular events ( MACE ) | during baseline to 6 months after therapy
  MACEs are defined as the occurrence of stroke, transient ischemic attacks (TIAs), blindness in patients.
The change value of arterial transit time ( ATT ) | during baseline to 6 months after therapy
  The change value of arterial transit time ( ATT ) in pCASL hypoperfusion area compared with baseline
The number of patients with erythema,and/or skin lesions related to RIC | during baseline to 6 months after therapy
  Professional doctors will check it and the investigator will record the number.
The number of patients with palpation for tenderness related to RIC | during baseline to 6 months after therapy
  Professional doctors will definite whether there's a palpation for tenderness and record the number.
The number of patients not tolerating RIC procedure,and refuse to continue the RIC procedure | during baseline to 6 months after therapy
  The investigator will record the number.
The number of patients with any other adverse events related to RIC intervention | during baseline to 6months after therapy
  The investigator will record the number.
Incidence of clinical symptoms | during baseline to 1, 2, 3, 6months after therapy
  The investigator will observe and record the occurrence of the clinical symptoms of dizziness, limb claudication, pulse deficits, bruits, headache, neck pain, severe abdominal pain, hypertension, valvular insufficiency, arrhythmia, chest pain or dsypnea.
The change value of blood pressure (BP) | during baseline to 1, 2, 3, 6months after therapy
  The change value of blood pressure (BP) will be compared with baseline
The change value of erythrocyte sedimentation rate (ESR) | during baseline to 1, 2, 3, 6months after therapy
  The change value of erythrocyte sedimentation rate (ESR) will be compared with baseline
The change value of C reactive protein (CRP) | during baseline to 1, 2, 3, 6months after therapy
  The change value of C reactive protein (CRP) will be compared with baseline
The change value of C reactive proteininterleukin 6 (IL-6) | during baseline to 1, 2, 3, 6months after therapy
  The change value of interleukin 6 (IL-6) will be compared with baseline
The change value of serum level of vascular endothelial growth factor (VEGF) | during baseline to 6months after therapy
  The change values of serum level of vascular endothelial growth factor (VEGF) will be compared with baseline.
The change value of serum level of nerve growth factor (NGF) | during baseline to 6months after therapy
  The change value of serum level of nerve growth factor (NGF) will be compared with baseline.
The change value of serum level of endothelin-1 (ET-1) | during baseline to 6months after therapy
  The change value of serum level of endothelin-1 (ET-1) will be compared with baseline.
The change value of serum level of angiotensin converting enzyme (ACE) | during baseline to 6months after therapy
  The change value of serum level of angiotensin converting enzyme (ACE) will be compared with baseline.
The change value of serum level of platelet activating factor (PAF) | during baseline to 6months after therapy
  The change value of serum level of platelet activating factor (PAF) will be compared with baseline.
The change value of serum level of platelet growth factor ( PDGF ) | during baseline to 6months after therapy
  The change value of serum level of platelet growth factor ( PDGF ) will be compared with baseline.
The change value of Birmingham Vasculitis Activity Score (BVAS) | during baseline to 6months after therapy
  The investigator will record the score. The BVAS is the most effective validated tool to document disease activity, ranging from 0 to 63. A score greater than or equal to 15 indicates that the disease is active. The higher score means the higher disease activity and a worse outcome.
The change value of the Indian Takayasu Clinical Activity Score (ITAS) 2010 | during baseline to 6months after therapy
  The investigator will record the score. ITAS 2010, a useful measure of clinical disease activity, ranges from 0 to 51 points. A score greater than or equal to 2 indicates that the disease is active. The higher score means the higher disease activity and the worse outcome.
The change value of the Vasculitis Damage Index (VDI) | during baseline to 6months after therapy
  Disease damage will be evaluated using the Vasculitis Damage Index (VDI). It ranges from 0 to 64 points. The higher score means the more severe vascular damage and the worse outcome.
The change value of the number of affected blood vessels | during baseline to 6months after therapy
  The number of affected blood vessels will be performed by Doppler US, CT angiography, magnetic resonance angiography (MRA), or digital subtraction angiography. The change value of the number will be compared with baseline.
Rate of the usage of glucocorticoids | during baseline to 6months after therapy
  The investigator will observe and record the usage of glucocorticoids.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Zhao, MD, Principal Investigator — Xuanwu Hospital, Capital Medical University, China, 10053; Sijie Li, MD, Principal Investigator — Xuanwu Hospital, Capital Medical University, China, 10053
Locations (1):
- Department of Rheumatology and Allergy, Xuanwu Hospital, Capital Medical University, Beijing, China, Beijing, Beijing Municipality, China